CLINICAL TRIAL: NCT01035567
Title: Prospective Randomised Pilot Study Evaluating the Safety and Efficacy of Hybrid Revascularization in Multivessel Coronary Artery Disease
Brief Title: Safety and Efficacy Study of Hybrid Revascularization in Multivessel Coronary Artery Disease
Acronym: POL-MIDES
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Silesian Centre for Heart Diseases (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Marian Zembala, MD, PhD, Head of the Cardiosurgery and Transplantology Department, Silesian Centre for Heart Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N R13 008406/2009
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Heart Disease; Myocardial Ischaemia; Coronary Disease; Coronary Artery Disease
Keywords: Multivessel coronary artery disease; Hybrid revascularization; Coronary Artery Bypass Grafting; Percutaneous Coronary Interventions; Drug eluting stents
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Coronary Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid revascularization (Active Comparator)
  Interventions: Procedure: Hybrid revascularization
- Coronary Artery Bypass Grafting (Active Comparator)
  Interventions: Procedure: Coronary Artery Bypass Grafting

INTERVENTIONS:
Procedure: Hybrid revascularization — First stage: implantation of the internal mammary artery into LAD in MIDCAB/TECAB procedure Second stage: PCI with drug eluting stents in other coronary arteries qualified for revascularization within 36 hours after surgery
  Arms: Hybrid revascularization
Procedure: Coronary Artery Bypass Grafting — Coronary artery bypass grafting with sternotomy on or off the pump at discretion of the operator.
  Arms: Coronary Artery Bypass Grafting

SUMMARY:
The purpose of the study is to assess the safety and efficacy of hybrid revascularization in comparison with coronary artery bypass grafting among patients with multivessel coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* Angiographically confirmed multivessel CAD with involved LAD and critical (>70%)lesion in at least one (apart LAD) major epicardial vessel amenable to both PCI and CABG
* Indication for revascularization based upon symptoms of angina and/or objective evidence of myocardial ischaemia
* Patient is willing to comply with all follow-up visits
* Patient signed an Informed Consent

Exclusion Criteria:

* Severe congestive heart failure (class III or IV according to NYHA, or pulmonary edema, cardiogenic shock) at the time of enrollment
* Prior surgery with the opening of pericardium or pleura
* Prior stroke (within 6 months)or more than 6 months if there are substantial neurological defects
* Prior history of significant bleeding (within previous 6 months) that might be expected to occur during PCI/CABG related anticoagulation
* One or more chronic total occlusions in major coronary territories
* Left main stenosis (at least 50% diameter stenosis)
* Acute ST-elevation MI within 72 hours prior to enrollment requiring revascularization
* Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stenting)
* Contraindication to either CABG, MIDCAB or PCI/DES because of a coexisting clinical condition
* Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis.
* Intolerance or contraindication to aspirin or both clopidogrel and ticlopidine
* Extra-cardiac illness that is expected to limit survival to less than 5 years e.g. oxygen-dependent chronic obstructive pulmonary disease, active hepatitis or significant hepatic failure, severe renal disease
* Suspected pregnancy. A pregnancy test will be administered prerandomization to all women of child-bearing age
* Concurrent enrollment in another clinical trial
* Patient inaccessible for follow-up visits required by protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-11; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Possibility defined by means of (1) a % of pts with complete hybrid procedure according to study protocol, and (2) a % of conversion to standard CABG. Safety defined as a occurrence of MACE such as death, MI, stroke, TVR, or major bleeding. | 1 year

SECONDARY OUTCOMES:
Postprocedure and follow up angiographic measurements as patency of grafts and restenosis in revascularized segments | 1 year
Assessment of quality of life of alive study participants according to SF-36 Health Survey version 2 | 1 year
Cost-effectiveness defined as a cost of revascularization procedure and costs of hospitalizations in both groups. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marian Zembala, PhD, Principal Investigator — Silesian Center for Heart Disease; Mariusz Gasior, PhD, Study Chair — Silesian Center for Heart Disease
Locations (2):
- Poland (2):
  - Department of Cardiosurgery and Transplatology, Silesian Medical University, Silesian Center for Heart Disease, Zabrze
  - Third Department of Cardiology, Silesian Medical University, Silesian Center for Heart Disease, Zabrze

REFERENCES:
- [Background] Riess FC, Schofer J, Kremer P, Riess AG, Bergmann H, Moshar S, Mathey D, Bleese N. Beating heart operations including hybrid revascularization: initial experiences. Ann Thorac Surg. 1998 Sep;66(3):1076-81. doi: 10.1016/s0003-4975(98)00714-0. PMID 9769007
- [Background] Wittwer T, Cremer J, Klima U, Wahlers T, Haverich A. Myocardial "hybrid" revascularization: intermediate results of an alternative approach to multivessel coronary artery disease. J Thorac Cardiovasc Surg. 1999 Oct;118(4):766-7. doi: 10.1016/S0022-5223(99)70035-8. No abstract available. PMID 10504652
- [Background] Cisowski M, Morawski W, Drzewiecki J, Kruczak W, Toczek K, Bis J, Bochenek A. Integrated minimally invasive direct coronary artery bypass grafting and angioplasty for coronary artery revascularization. Eur J Cardiothorac Surg. 2002 Aug;22(2):261-5. doi: 10.1016/s1010-7940(02)00262-2. PMID 12142196
- [Background] Stahl KD, Boyd WD, Vassiliades TA, Karamanoukian HL. Hybrid robotic coronary artery surgery and angioplasty in multivessel coronary artery disease. Ann Thorac Surg. 2002 Oct;74(4):S1358-62. doi: 10.1016/s0003-4975(02)03889-4. PMID 12400817
- [Derived] Tajstra M, Hrapkowicz T, Hawranek M, Filipiak K, Gierlotka M, Zembala M, Gasior M, Zembala MO; POL-MIDES Study Investigators. Hybrid Coronary Revascularization in Selected Patients With Multivessel Disease: 5-Year Clinical Outcomes of the Prospective Randomized Pilot Study. JACC Cardiovasc Interv. 2018 May 14;11(9):847-852. doi: 10.1016/j.jcin.2018.01.271. Epub 2018 Apr 18. PMID 29680218
- [Derived] Gasior M, Zembala MO, Tajstra M, Filipiak K, Gierlotka M, Hrapkowicz T, Hawranek M, Polonski L, Zembala M; POL-MIDES (HYBRID) Study Investigators. Hybrid revascularization for multivessel coronary artery disease. JACC Cardiovasc Interv. 2014 Nov;7(11):1277-83. doi: 10.1016/j.jcin.2014.05.025. Epub 2014 Nov 17. PMID 25459040
- [Derived] Zembala M, Tajstra M, Zembala M, Filipiak K, Knapik P, Hrapkowicz T, Gierlotka M, Hawranek M, Polonski L, Gasior M. Prospective randomised pilOt study evaLuating the safety and efficacy of hybrid revascularisation in MultI-vessel coronary artery DisEaSe (POLMIDES) - study design. Kardiol Pol. 2011;69(5):460-6. PMID 21594832